CLINICAL TRIAL: NCT01789229
Title: Establishment of a Tissue Sample Bank in the Field of Gynaecological Oncology
Brief Title: Establishment of a Tumor Bank for Tissue Samples
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Robert Zeillinger, Dr.phil., Univ.Prof. Dr., Medical University of Vienna
Other Study IDs: EK 260/2003
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Neoplasms of the Female Genitalia; Lung Neoplasms; Endocrine Gland Neoplasms
Keywords: biobank; fresh-frozen tissue
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Endocrine Gland Neoplasms | interventions — Therapeutic Irrigation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Universal tumor bank
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Malignant tumors: Patients who have one of the Neoplasms stated above under "conditions".
  Interventions: Other: Tumor tissue collection; Other: Sampling of ascites and pleural effusion; Other: Collecting urine samples; Other: Collecting saliva sample; Other: Collecting sputum; Other: Collecting stool samples; Other: Lavage/Irrigation
- Benign controls: Patients with a benign tumor or an inflammatory disease - to be matched by age.
  Interventions: Other: Tumor tissue collection; Other: Sampling of ascites and pleural effusion; Other: Collecting urine samples; Other: Collecting saliva sample; Other: Collecting sputum; Other: Collecting stool samples; Other: Lavage/Irrigation
- Healthy controls: People/patients who have no known disease at time of sampling or are admitted to the hospital for minor interventions and have no inflammatory disease.
  Interventions: Other: Collecting urine samples; Other: Collecting saliva sample; Other: Collecting sputum; Other: Collecting stool samples; Other: Lavage/Irrigation

INTERVENTIONS:
Other: Tumor tissue collection — Tissue sample is collected during therapeutic intervention by a medical doctor/surgeon.
  Frozen tissue sections are first transferred to Dept.of Pathology. Pathologist samples required tissue to obtain enough evidence for analysis/diagnosis.
  Rest tumor material with or without malignant cells is tranferred to the lab for Molecular Oncology of Prof.Zeillinger.
  Groups: Benign controls; Malignant tumors
Other: Sampling of ascites and pleural effusion — Samples of malignant ascites and/or malignant pleural effusion is only collected during therapeutic intervention from patients at inpatient care.
  Groups: Benign controls; Malignant tumors
Other: Collecting urine samples — Patient is asked to give a urine sample. Urine is collected in urine beaker.
Other: Collecting saliva sample — Saliva sample is collected by spatula from the mouth cavity of the patient.
Other: Collecting sputum — Patient is asked to produce sputum into a 50ml lab tube.
Other: Collecting stool samples — Stool samples are collected prior to bowel preparation for colonoscopy. Device for sampling is provided to the patient.
Other: Lavage/Irrigation — Irrigation liquid is collected during routine therapeutic or diagnostic procedure, e.g. lavage of the uterine cavity and fallopian tubes of women scheduled for surgery.

SUMMARY:
Establishment of a tumor bank, consisting of tissue samples of tumor patients (benign and malign tumors) and healthy people as controls. The tissue samples will be collected systematically together with the corresponding clinical data. The biological samples, the clinical date together with prospective experimental date constitute the entity of the tissue tumor bank.

This tumor bank for tissue samples, together with our tumorbank for blood samples (NCT01763125) combined constitute the entity "Tumorbank".

DETAILED DESCRIPTION:
Recent progress in diagnosis and therapy of cancer diseases can be ascribed mainly to translational research. The relevance of "translational oncology" will only increase in the future -"From bench to bedside" - the swift implementation of new science research results in clinical studies in order to expedite progress in clinical cancer therapy for the benefit of the patient.

Its almost a matter of course in the medical science today to collect biological samples together with clinical information thereby creating the foundation for future excellent fundamental research.

The aim of this tumor bank is to consist of biological samples (together with a blood bank - see NCT01763125) and isolates of tumor patients and healthy people as controls. The biological samples, the clinical date together with prospective experimental date constitute the entity of the tumor bank. The content of the tumor bank can provide essential material for current and future research (e.g. analyses of prognostic or predictive tumor markers; genetically analysis (polymorphism, mutation, hypermethylation; verification and characterisation of disseminated tumor cells).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Age 18 to 90 years max.
* Just one current known malignant disease or just one current inflammatory disease

Exclusion Criteria:

* Inflammatory disease and malignant disease
* multiple malignancies
* multiple diseases
* underage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients/people. Minimum age 18 years Characteristics: Recruited at the Medical University Vienna or at one of the facilities cooperating with the Vienna Med. University
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2003-09; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Establishment of blood/tissue bank consisting of oncological samples from cancer patients and benign and healthy controls. | 14 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeillinger, Prof.Dr., Principal Investigator — Medical University of Vienna, Dptm. of Obstetrics & Gynaecology
Locations (3):
- Medical University Vienna, Dptm. of Obstetrics & Gynaecology, Vienna, Austria
- University Hospitals Leuven - Department of Obstetrics and Gynaecology, Leuven, Belgium
- Charité University - Campus Virchow Chlinic, Berlin, Germany

REFERENCES:
- [Result] Hofstetter G, Berger A, Fiegl H, Slade N, Zoric A, Holzer B, Schuster E, Mobus VJ, Reimer D, Daxenbichler G, Marth C, Zeimet AG, Concin N, Zeillinger R. Alternative splicing of p53 and p73: the novel p53 splice variant p53delta is an independent prognostic marker in ovarian cancer. Oncogene. 2010 Apr 1;29(13):1997-2004. doi: 10.1038/onc.2009.482. Epub 2010 Jan 18. PMID 20101229
- [Result] Tong D, Heinze G, Pils D, Wolf A, Singer CF, Concin N, Hofstetter G, Schiebel I, Rudas M, Zeillinger R. Gene expression of PMP22 is an independent prognostic factor for disease-free and overall survival in breast cancer patients. BMC Cancer. 2010 Dec 15;10:682. doi: 10.1186/1471-2407-10-682. PMID 21159173
- [Result] Grimm C, Watrowski R, Baumuhlner K, Natter C, Tong D, Wolf A, Zeillinger R, Leodolter S, Reinthaller A, Hefler L. Genetic variations of interleukin-1 and -6 genes and risk of cervical intraepithelial neoplasia. Gynecol Oncol. 2011 Jun 1;121(3):537-41. doi: 10.1016/j.ygyno.2011.02.019. Epub 2011 Mar 3. PMID 21376376
- [Result] Hofstetter G, Berger A, Schuster E, Wolf A, Hager G, Vergote I, Cadron I, Sehouli J, Braicu EI, Mahner S, Speiser P, Marth C, Zeimet AG, Ulmer H, Zeillinger R, Concin N. Delta133p53 is an independent prognostic marker in p53 mutant advanced serous ovarian cancer. Br J Cancer. 2011 Nov 8;105(10):1593-9. doi: 10.1038/bjc.2011.433. Epub 2011 Oct 18. PMID 22009029
- [Result] Pils D, Horak P, Vanhara P, Anees M, Petz M, Alfanz A, Gugerell A, Wittinger M, Gleiss A, Auner V, Tong D, Zeillinger R, Braicu EI, Sehouli J, Krainer M. Methylation status of TUSC3 is a prognostic factor in ovarian cancer. Cancer. 2013 Mar 1;119(5):946-54. doi: 10.1002/cncr.27850. Epub 2012 Oct 23. PMID 23096450